CLINICAL TRIAL: NCT00557921
Title: A Randomized, Double-Blind, Double-Dummy, Parallel Group, Phase 3 Efficacy and Safety Study of CGT-2168 Compared With Clopidogrel to Reduce Upper Gastrointestinal Events Including Bleeding and Symptomatic Ulcer Disease
Brief Title: Clopidogrel and the Optimization of Gastrointestinal Events (COGENT-1)
Acronym: COGENT-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Cogentus Pharmaceuticals (Industry)
Responsible Party: Pablo Lapuerta, MD, Cogentus Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CG104; EudraCT 2007-005891-15
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: ACS; CAD; MI; PCI; PTCA; NSTEMI; STEMI; acute coronary syndrome; cerebrovascular disorders; coronary artery stent placement; coronary thrombosis; myocardial infarction; myocardial ischemia; percutaneous coronary intervention; percutaneous transluminal coronary angioplasty; peripheral vascular diseases; duodenal obstruction; duodenal ulcer; dyspepsia; esophagitis, peptic; gastric outlet obstruction; gastroduodenal ulcer; gastroesophageal reflux disease; gastrointestinal hemorrhage; peptic ulcer; peptic ulcer perforation
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Coronary Artery Disease; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Cerebrovascular Disorders; Coronary Thrombosis; Myocardial Ischemia; Peripheral Vascular Diseases; Duodenal Obstruction; Duodenal Ulcer; Dyspepsia; Esophagitis, Peptic; Gastric Outlet Obstruction; Peptic Ulcer; Gastroesophageal Reflux; Gastrointestinal Hemorrhage; Peptic Ulcer Perforation | interventions — Clopidogrel; Omeprazole; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CGT-2168 (clopidogrel 75 mg/omeprazole 20 mg) and aspirin
- 2 (Active Comparator)
  Interventions: Drug: Plavix (clopidogrel 75 mg) and aspirin

INTERVENTIONS:
Drug: CGT-2168 (clopidogrel 75 mg/omeprazole 20 mg) and aspirin — (CGT-2168 active and Comparator placebo, one capsule each daily; and enteric coated aspirin at daily dose level assigned by study physician)
  Arms: 1
Drug: Plavix (clopidogrel 75 mg) and aspirin — (CGT-2168 placebo and Comparator active, one capsule each daily; and enteric coated aspirin at daily dose level assigned by study physician)
  Arms: 2

SUMMARY:
The purpose of the COGENT-1 clinical trial is to determine whether CGT-2168 (clopidogrel and omeprazole) compared to clopidogrel is safe and effective in reducing the incidence of gastrointestinal bleeding and symptomatic ulcer disease, in the setting of concomitant aspirin therapy.

Antiplatelet therapy is an essential element of care for patients with atherothrombotic disease. Bleeding is a fundamental adverse effect of all antiplatelet drugs including aspirin, clopidogrel and dual antiplatelet regimens.

The gastrointestinal tract is the most common site of bleeding related to antiplatelet therapy, typically in connection with peptic ulcer disease. Recently published studies suggest the use of clopidogrel carries a gastrointestinal bleeding risk similar to that of aspirin or non-aspirin non-steroidal anti-inflammatory drugs. Patients taking any two of these drugs (clopidogrel, aspirin and/or non-aspirin NSAIDs) are exposed to an even higher risk of bleeding and ulcer disease.

Cogentus Pharmaceuticals is launching phase 3 trials of a novel combination product, CGT-2168, which has the potential to significantly reduce this problem and increase patient safety. CGT-2168 combines a standard dosage of clopidogrel and a gastroprotectant (omeprazole) in a once-daily pill that may reduce the likelihood of adverse gastrointestinal events.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom a requirement for clopidogrel therapy with concomitant aspirin is anticipated for at least the next 12 months. Specific conditions that may confer a need for long-term clopidogrel + aspirin therapy may include non-ST segment elevation acute coronary syndrome (unstable angina/non-Q-wave MI), ST segment elevation acute MI), or new placement of a coronary artery stent.
* For women of childbearing potential, negative pregnancy test prior to randomization and agreement to use effective method of birth control during the study.
* Able to provide written informed consent based on competent mental status.

Exclusion Criteria:

* Patients currently hospitalized for whom discharge is not anticipated within 48 hours of randomization.
* Requirement for current or chronic use of a proton pump inhibitor, H2 receptor blocker, sucralfate or misoprostol.
* Erosive esophagitis, esophageal or gastric variceal disease, or non-endoscopic gastric surgery. Patients with a history of GERD/erosive esophagitis or dyspepsia who do not currently require proton pump blockers will be eligible.
* Receipt of > 21 days of clopidogrel or another thienopyridine prior to randomization.
* Oral anticoagulation that cannot be safely discontinued for duration of study.
* Recent fibrinolytic therapy.
* Scheduled percutaneous coronary intervention (PCI). Patients may be enrolled upon completion of PCI.
* Recent (< 30 days prior to randomization) or scheduled coronary artery bypass graft (CABG) surgery.
* Cardiogenic shock at time of randomization, refractory ventricular arrhythmias, or congestive heart failure (NY Heart Association class IV).
* Active pathological bleeding or a history of hereditary or acquired hemostatic disorder.
* History of hemorrhagic stroke, intracranial neoplasm, arteriovenous malformation or aneurysm.
* Systemic corticosteroids except low-dose oral corticosteroids equivalent to prednisone < or equal to 5 mg/day.
* Allergy or contraindication to clopidogrel or other thienopyridine drugs, omeprazole or other proton pump inhibitor drugs, aspirin or salicylate derivatives, or other study drug ingredients.
* Treatment within 30 days prior to randomization with any investigational drug or device including investigational coronary artery stents or currently enrolled in another interventional drug or device study.
* Women who are pregnant or breastfeeding.
* Life expectancy less than 12 months.
* Laboratory abnormality at screening that is clinically significant or outside protocol-allowed limits, or any other condition that precludes participation in the study in the opinion of the Investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Composite of upper gastrointestinal clinical events, including gastroduodenal bleeding, symptomatic gastroduodenal ulcer, persistent pain with multiple gastric erosions, obstruction or perforation | Anticipated minimum of 48 weeks, up to end of study

SECONDARY OUTCOMES:
Composite of gastroduodenal bleeding, symptomatic gastroduodenal ulcer, obstruction or perforation | Anticipated minimum of 48 weeks, up to end of study
Composite of gastroduodenal bleeding, obstruction or perforation | Anticipated minimum of 48 weeks, up to end of study
Discontinuation of study medication attributed to gastrointestinal signs or symptoms | Anticipated minimum of 48 weeks, up to end of study
Gastroesophageal reflux disease, as evidenced by symptomatic endoscopically-confirmed erosive esophagitis | Anticipated minimum of 48 weeks, up to end of study
Dyspepsia, defined as an increase of at least ten points on the "pain intensity" component of the SODA instrument from baseline | Anticipated minimum of 48 weeks, up to end of study
Occurrence of a cardiovascular event (cardiovascular death, nonfatal myocardial infarction, CABG or PCI, or confirmed ischemic stroke | Anticipated minimum of 48 weeks, up to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Lapuerta, MD, Study Director — Cogentus Pharmaceuticals
Locations (487):
- United States (243):
  - Alabama Clinical Research Institute, Inc. (ACRI), Alexander City, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Cardio-Thoracic Surgeons P.C., Birmingham, Alabama
  - Birmingham Heart Clinic, PC, Birmingham, Alabama
  - John F Simmons , MD PC, Geneva, Alabama
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - The Heart Center, PC, Huntsville, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Advanced Cardiac Specialists, Mesa, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Cardiovascular Consultants, Ltd., Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Paradigm Clinical Research, Inc., Tucson, Arizona
  - Tri-Lakes Research, Hot Springs, Arkansas
  - Michael A. Frais, Cardiologist, P.A., Hot Springs, Arkansas
  - NEA-Clinic Cardiology, Jonesboro, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - Cardiology Consultants of Orange County, Anaheim, California
  - Chest and Critical Care Consultants, A Medical Group, Anaheim, California
  - Clinical Solutions Advantage, Buena Park, California
  - Turns Institute for Clinical Research, Castro Valley, California
  - Escondido Cardiology Associates, Escondido, California
  - Accurate Clinical Trials, Inc., Laguna Hills, California
  - Therapeutic Research Institute of Orange County, Laguna Hills, California
  - Kirtik Thaker MD, Lakewood, California
  - Los Angeles Cardiology Associates, Los Angeles, California
  - Merced Heart Associates, Merced, California
  - Mission Internal Medical Group, Mission Viejo, California
  - Altos Cardiovascular Associates, Mountain View, California
  - Kenneth W. Carr, MD, Cardiology, Oceanside, California
  - Rancho CucamongaClinical Trials, Rancho Cucamonga, California
  - Inland Heart and Vascular Medical Associates, San Bernardino, California
  - Ritchken and First, San Diego, California
  - Rider Research Group, San Francisco, California
  - Richard Levy, MD., San Francisco, California
  - Kaiser Permanente, San Jose, California
  - Medical Helping Hands Research, Santa Ana, California
  - Pacific Heart Institute, Santa Monica, California
  - Radiant Research, Santa Rosa, California
  - Harbor- UCLA Medical Center, Torrance, California
  - Ventura Cardiology Consultants Medical Group, Inc., Ventura, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Connecticut Clinical Research, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Alfieri Cardiology, PA, Newark, Delaware
  - Washington V.A. Medical Center, Washington D.C., District of Columbia
  - Oscar R. Guerra, MD PA, Coral Gables, Florida
  - Deerfield Beach Cardiology Associates, Deerfield Beach, Florida
  - Dr Jules Cohen, Hallandale, Florida
  - Empire International Research, Hialeah, Florida
  - Cardiovascular Consultants of South Florida, Hollywood, Florida
  - Jacksonville Heart Center, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - CVMS Resesarch Institute, LLC, Jupiter, Florida
  - Watson Clinic Center for Research, Lakeland, Florida
  - Alpha Medical Research, LLC, Melbourne, Florida
  - Empire International Research, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Research Center Phase I-IV of Florida Corp., Miami, Florida
  - Bert Fish Medical Center, New Smyrna Beach, Florida
  - Central Florida Cardiology Group, Orlando, Florida
  - Cardiology Assocaites of Orlando d/b/a Orlando Heart Center, Orlando, Florida
  - Sunset Point Medical Associates, Palm Harbor, Florida
  - Berma Research Group, Plantation, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Suncoast Cardiovascular Research, St. Petersburg, Florida
  - The Heart and Vascular Institute of Florida, St. Petersburg, Florida
  - G&G Research Baker-Tombul Cardiology, Vero Beach, Florida
  - Carlos Levy, D.O., Weston, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Primary Care Specialists, LLC/ ECAST CT, Atlanta, Georgia
  - Executive Health and Research Associates, Inc., Atlanta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Georgia Heart Specialists, LLC, Covington, Georgia
  - Ialum Clinical Research Center, LLC, Decatur, Georgia
  - Ialum Clinical Research Center, Decatur, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - Medsouth Primary CareStockbridge, Stockbridge, Georgia
  - South Suburban Health Professional Group, PC, Flossmoor, Illinois
  - Consultants in Cardiovascular Medicine, Melrose Park, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - American Health Network, Avon, Indiana
  - Indiana Medical Research, Elkhart, Indiana
  - Welborn Clinic, Evansville, Indiana
  - Indiana Heart Physicians, Indianapolis, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - Hutchinson Clinic, P.A., Hutchinson, Kansas
  - Venture Resource Group, Inc., Mission, Kansas
  - Midwest Cardiology Assocaites, Overland Park, Kansas
  - Cumberland Cardiology, Ashland, Kentucky
  - Trover Health System, Madisonville, Kentucky
  - Owensboro Heart and Vascular, Owensboro, Kentucky
  - Dolby Research, LLC, Baton Rouge, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Heart Clinic of Louisiana Clinical Research, LLC., Marrero, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Cardiovascular Consultants of Maine, PA, Scarborough, Maine
  - Maine Cardiology Associates, South Portland, Maine
  - Good Samaritan Hospital (Medstar Health), Baltimore, Maryland
  - eCast Corporation, Greenbelt, Maryland
  - Atlantic Cardiology Associates, P.A, Salisbury, Maryland
  - Peninsula Cardiology Associates, Salisbury, Maryland
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Michigan Cardiovascular Institute, Bay City, Michigan
  - Apex Medical Research, AMR, Inc., Flint, Michigan
  - Borgess Research Institute, Kalamazoo, Michigan
  - Michigan Cardiovascular Institute, Midland, Michigan
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Academic Heart and Vascular PLLC, Saint Clair Shores, Michigan
  - Oakland Medical Center, Troy, Michigan
  - Waterford Medical Assoc. P.C., Waterford, Michigan
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Duluth Clinic / Saint Marys Medical Center, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - New Coast Cardiology Center, PLLC, Gulfport, Mississippi
  - PPS Clinical Research, STL, LLC, Chesterfield, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Cardiology Diagnostics, Ltd., St Louis, Missouri
  - Glacier View Cardiology, Kalispell, Montana
  - Saint Patrick Hospital- International Heart Institute of Montana, Missoula, Montana
  - The Creighton Cardiac Center, Omaha, Nebraska
  - Alegent Health Clinic Heart and Vascular Specialist, Papillion, Nebraska
  - Nevada Cardiology Associates, Las Vegas, Nevada
  - Lahey Cardiology @ the Medical Center, Nashua, New Hampshire
  - Associated Cardiovascular Consultants, Cherry Hill, New Jersey
  - Cardiovascular Associates of the Delaware Valley, P.A., Elmer, New Jersey
  - Cardiovascular Associates of the Delaware Valley, P.A., Haddon Heights, New Jersey
  - Cardiovascular Associates of the Delaware Valley, P.A., Sewell, New Jersey
  - Physicans Research Center, LLC, Toms River, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - Hudson Valley Cardiology Group, P.C., Cortlandt Manor, New York
  - Cardiology Associates, P.C., Johnson City, New York
  - Long Island Heart Associates, Mineola, New York
  - Slocum-Dickson Medical Group, PLLC, New Hartford, New York
  - Sound Shore Cardiology, P.C., New Rochelle, New York
  - New York Cardiovascular Associate, New York, New York
  - St. Luke's- Roosevelt Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Saratoga Cardiology Assoc, PC, Saratoga Springs, New York
  - Westchester Cardiology Associates, Scarsdale, New York
  - Good Samaritan Hospital, Suffern, New York
  - Cardiology, PC, Syracuse, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cardiac Care and Vascular Medicine, Albert Einstein College of Medicine, The Bronx, New York
  - Capital Cardiology Associates, Troy, New York
  - Buffalo Cardiology and Pulmonary Associates, Williamsville, New York
  - Mark J. Kozinn, MD, Williamsville, New York
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Kernodle Clinic, Inc., Burlington, North Carolina
  - Metrolina Medical Research, Charlotte, North Carolina
  - Diversified Research, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Cardiovascular Care of Northern Carolina, Oxford, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - Trinity Health, Minot, North Dakota
  - George G. Ellis, Jr. M.D., Inc., Boardman, Ohio
  - Cardiovascular Research Institute, LLC, Canton, Ohio
  - Comprehensive Cardiology Consultants, Inc., Cincinnati, Ohio
  - Midwest Cardiology Research Foundation, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Cardiology Associates of SE Ohio, Inc, Zanesville, Ohio
  - Physicans Research, Inc., Zanesville, Ohio
  - Bluestem Cardiology Research Dept., Bartlesville, Oklahoma
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Aquilo Research, Yukon, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Hillsboro Cardiology, PC, Hillsboro, Oregon
  - Legacy Clinical Research, Portland, Oregon
  - Abington Medical Specialists, Abington, Pennsylvania
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Heritage Cardiology Association, Camp Hill, Pennsylvania
  - Premier Heart Specialists, Easton, Pennsylvania
  - Heart Specialists of Lancaster, Ephrata, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Pennsylvania Heart and Vascular Group, P.C., Jenkintown, Pennsylvania
  - Comprehensive Cardiology Consultants, Langhorne, Pennsylvania
  - Sewickley Valley Medical Group Cardiology, Leetsdale, Pennsylvania
  - Cardiology Consultants of Philadelphia, Norristown, Pennsylvania
  - Hospital of the University of Pennsylvania Cardiology Department, Philadelphia, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Advanced Cardiology Specialists, Scranton, Pennsylvania
  - Elite Medical Research, Inc., Sellersville, Pennsylvania
  - Cardiology Consultants of Philadelphia, Upland, Pennsylvania
  - West Chester Cardiology, PC, West Chester, Pennsylvania
  - Berks Cardiology, Ltd., Wyomissing, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - New England Center for Clinical Research&comma; Inc, Cranston, Rhode Island
  - Rhode Island Hospital Cardiology, Providence, Rhode Island
  - Cardiology Specialists, Westerly, Rhode Island
  - Palmetto Clinical Research, Summerville, South Carolina
  - McMinn Medical Group (DBA: Athens Medical Group), Athens, Tennessee
  - Verzosa & Ungab Internal Medicine Associates, Bartlett, Tennessee
  - Middle Tennessee Clinical Research, Fayetteville, Tennessee
  - Research Associates of Jackson and Apex Cardiology, Jackson, Tennessee
  - Tri-State Cardiology, Johnson City, Tennessee
  - Memphis Internal Medicine, Memphis, Tennessee
  - Goodlife Medical Center, Memphis, Tennessee
  - Heart and Vascular Clinic, Nashville, Tennessee
  - Family Health Care Assoc., Arlington, Texas
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Trinity Hypertension and Diagnostic Res., Carrollton, Texas
  - VA Medical Center, Dallas, Texas
  - U.T. Southwestern, Dallas, Texas
  - Amir Malik Research, Fort Worth, Texas
  - The University of Texas Medical Branch at Galveston, Galveston, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Office of Amer Zaheer, MD, Houston, Texas
  - Office of Salim Gopalani, MD, Houston, Texas
  - Comprehensive Heart Care, PA, Houston, Texas
  - Century Clinical Research, Houston, Texas
  - Office of Mizra Basith Baig, MD, Houston, Texas
  - Covenant Cardiology Associates, Lubbock, Texas
  - South Texas Institutes of Health, McAllen, Texas
  - Texas Regional Heart Center d/b/a Legacy Heart Center, Plano, Texas
  - Heart & Vascular Institute of Texas, San Antonio, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - IMED Research, PA, San Antonio, Texas
  - Southwest Health Associate, PA, Sugar Land, Texas
  - Office of Dwayne O. Williams, MD, Sugarland, Texas
  - Kings Daughters Clinic, Temple, Texas
  - Victoria Heart and Vascular Center, Victoria, Texas
  - Cardiology Consultants of Danville, Danville, Virginia
  - Triad Research Institute, Galax, Virginia
  - Virginia Cardiovascular Specialists, Richmond, Virginia
  - Winchester Medical Center/ Clinical Research Department, Winchester, Virginia
  - Daniel W. Gottlieb, MD, PS, Burien, Washington
  - Heart Clinic Northwest, Spokane, Washington
  - Inland Cardiology Assocaites, Spokane, Washington
  - Franciscan Health System dba FHS Research Center, Tacoma, Washington
  - Parkersburg Cardiology Associates, Parkersburg, West Virginia
  - Wisconsin Heart, S.C., Madison, Wisconsin
  - Heart Care Associates, LLC, Milwaukee, Wisconsin
- Australia (12):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Coffs Harbour Cardiology, Coffs Harbour, New South Wales
  - Cardiac Research Institute, Eastwood, New South Wales
  - Wesley research institute, Auchenflower, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Northern Hospital, Epping, Victoria
  - St.Vincent's Hospital (Melb), Fitzroy, Victoria
  - Geelong Hospital- Barwon Health, Geelong, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
- Bulgaria (13):
  - Multiprofile Hospital for Active Treatment "Sveta Ekaterina", 1st Department of Internal Diseases, Dimitrovgrad
  - Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski, Clinic of Cardiology, Pleven
  - Multiprofile Hospital for Active Treatment ''Sveti Georgi'', Cardiology Clinic, Plovdiv
  - Multiprofile Hospital for Active Treatment ''Sveti Panteleymon'', 2nd Department. of Internal Diseases - Intensive Cardiology Unit, Plovdiv
  - Multiprofile Hospital for Active Treatment - Ruse, 4th Department of Internal Diseases, Rousse
  - 4th Multiprofile Hospital for Active Treatment, Sofia
  - Military Medical Academy, Clinic of Cardiology and Intensive Care, Sofia
  - Multiprofile Hospital for Active Treatment and Emergency Medicine "Pirogov". Cardiology Clinic, Sofia
  - National Heart Hospital Department of Cardiology, Sofia
  - National Multiprofile Transport Hospital "Tsar Boris III, Cardiology Clinic, Sofia
  - Tokuda Hospital Department of Cardiology, Sofia
  - University Multiprofile Hospital for Active Treatment ''Tsaritsa Ioanna'' - ISUL, Cardiology Clinic, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina", Clinic of Internal Diseases - 2nd Internal Department, Varna
- Canada (24):
  - Dr. Tsui, Maple Ridge, British Columbia
  - Fraser Clinical Trials Inc and Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - South East Regional Health Authority, Moncton, New Brunswick
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Mississauga Clinical Research Center, Mississauga, Ontario
  - Dr. George Zimakas, Niagara Falls, Ontario
  - Dr. James Y. Cha, Oshawa, Ontario
  - Curans Health Center, Thunder Bay, Ontario
  - Toronto East Cardiology Associates Inc., Toronto, Ontario
  - Recherches Cliniques Theradev, Granby, Quebec
  - ViaCar Recherche Clinique Inc., Greenfield Park, Quebec
  - ViaCar Recherche Clinique Inc, Longueuil, Quebec
  - Hospitalier de l'Universite de Montreal Hotel Dieu, Montreal, Quebec
  - Sacre-Coeur Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec (CHOQ) Hotel Dieu de Quebec, Québec, Quebec
  - Laval Hospital, Québec, Quebec
  - Centre Hospitalier Beauce-Etchemin, Saint George, Quebec
  - Centre de Sante et de services sociaux du nord de lanaudiere/CHRDL, Saint-Charles-Borromée, Quebec
  - Clinique de Cardiologie de Trois-Rivieres, Trois-Rivières, Quebec
  - Cardiology and Research, Westmount, Quebec
- Chile (10):
  - Clinica Antofagasta, Antofagasta
  - Corporación de Beneficencia Osorno, Osorno
  - Hospital Regional de Punta Arenas Dr. Lautaro Navarro, Punta Arenas
  - Complejo Asistencial Dr.Sótero del Río, Santiago
  - Hospital del Salvador, Santiago
  - Instituto Nacional del Tórax, Santiago
  - Centro de Estudios Cardiovascular, Temuco
  - Clínica Reñaca, Viña del Mar
  - Hospital Dr. Gustavo Fricke, Viña del Mar
  - Hospital Naval Almirante Neff, Viña del Mar
- Czechia (11):
  - Nemocnice ve Frydku-Mistku, Frýdek-Místek
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Krajska nemocnice Liberec, a. s., Liberec
  - Litomyslska nemocnice a. s., Litomyšl
  - Kardiologická ambulance, Ostrava
  - Kardiologicka a angiologicka ambulance, Ostrava Vítkovice
  - Pardubicka krajska nemocnice, a.s., Pardubice
  - II.interni klinika kardiologie a angiologie 1. LF UK a VFN v Praze, Prague
  - Klinika kardiologie Institut klinické a experimentální medicíny, Prague
  - Krajská nemocnice T. Bati a.s., Zlín
  - Nemocnice Znojmo, p.o., Znojmo
- France (9):
  - Centre Hospitalier d'Albi, Albi
  - Centre de Cardiologie CHRU Dijon, Dijon
  - Clinique Pasteur, Essey-lès-Nancy
  - CHRU de Lille Hôpital Cardiologique, Lille
  - Hôpital La Timone-Adultes, Marseille
  - Hôpital Lariboisière, Paris
  - La Pitié Salpétrière Institut de Cardiologie, Paris
  - Centre Hospitalier Intercommunal du Val d'Ariège, Saint-Jean-de-Verges
  - Centre Hospitalier Rangueil Larrey, Toulouse
- Germany (50):
  - Universitatsklinikum Berlin Campus Charite Mitte Med Klinik Kardiologie und Angiologie, Berlin
  - Vivantes Clinic Neuköln Berlin, Berlin
  - Vivantes Humbolt Klinikum, Berlin
  - Praxis Dr. med. Boscher, Biberach
  - St. Josef-Hospital Medizinische Klinik II, Kardiologie, Bochum
  - St.-Marien-Hospital Bonn, Bonn
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - MVZ am Küchwald GmbH, Chemnitz
  - Kliniken der Stadt Köln, Köln Merheim, Cologne
  - Gemeinschaftspraxis Innere Medizin und Kardiologie, Dinslaken
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden Neustadt GbR, Dresden
  - Practice of Cardiology, Erfurt
  - Elisabeth.Krankenhaus, Essen
  - Asklepios Klinik St.Georg, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Universitäres Herz-und Gefäßzentrum Hamburg", Hamburg
  - Kardiologische Praxis Hamburg Altona, Hamburg
  - Klinikum Region Hannover Krankenhaus Nordstadt, Hanover
  - Kardiologische Gemeinschaftspraxis, Hartmannsdorf
  - SRH Klinikum Karlsbad-Langensteinbach, Karlsbad
  - Herzzentrum Lahr, Lahr
  - Kardiologische Gemeinschaftpraxis, Leipzig
  - Universität Leipzig - Herzzentrum, Leipzig
  - Dr. THomas Klingenheben, Lengsdorf
  - Praxis für Innere Medizin, Gastroenterologie, Ludwigshafen
  - Universitätsklinikum Lübeck, Lübeck
  - Gemeinschaftspraxis, Lüneburg
  - Klinikum der Johannes-Gutenberg-Universität, Mainz
  - Gemeinschaftspraxis, Mannheim
  - Klinikum Mannheim GmbH, Universaitatskinikum, Mannheim
  - Kardiologische Praxis, Markkleeberg
  - Asklepios Klinik Melsungen, Melsungen
  - Kilniken Maria Hilf GmbH Krankenhaus St. Franziskus, Mönchengladbach
  - Internist/Kardiologe/Angiologe, Mühldorf A.d. Inn
  - Kardiologische Gemeinschaftspraxis, Nienburg
  - Klinikum Pirna GmbH, Pirna
  - Universitätsklinik Regensburg, Regensburg
  - Krankenhaus Reinbek St. Adolf-Stift, Reinbek
  - Kardiologische Gemeinschaftspraxis, Riesa
  - Internistische Praxis, Rottweil
  - Zentrum für Prävention und Rehabilation, Siegen
  - Marienkrankenhaus Soest, Soest
  - Praxisgemeinschaft Stuhr-Brinkum, Stuhr
  - Medizinische Universitätsklinik, Tübingen
  - Josephs-Hospital Warendorf, Warendorf
  - Kardiologische Praxis, Wermsdorf
  - Dr. Andreas Schreckenberg, Weyhe-Leeste
  - ForschungsZentrum Ruhr, Witten
  - Helios Klinikum Wuppertal, Wuppertal
- Hungary (9):
  - Bajai Kórház, Baja
  - Budai Irgalmasrendi Kórház, Budapest
  - Fővárosi Önkormányzat Károlyi Sándor Kórház és Rendelőintézet, Budapest
  - Fovarosi Onkormanyzat Egyesitett Szent Istvan es Szent Laszlo Korhaz - Rendelointezet, Budapest
  - Városi Önkormányzat Kórház-Rendelőintézet, Kalocsa
  - Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András Oktató Kórház, Nyíregyháza
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház, Toszegi
  - Jávorszky Ödön Kórház, Vác
  - Zala Megyei Kórház, Zalaegerszeg
- Italy (6):
  - Ospedali Riuniti di bergamo, Bergamo
  - Azienda Ospedaliera della Provincia di Lodi Presidio Ospedaliero di Codogno, Codogno (Lodi)
  - Azienda Ospedaliera Universitaria San Martino-Dipartimento di Medicina Interna e Specialità Mediche, Genova
  - Azienda Ospeedaliera Carlo Poma, Mantova
  - Azienda Ospedaliera Maggiore Della Carita' Di Novara, Novara
  - Istituto Clinico Humanitas, Rozzano (Milano)
- Mexico (9):
  - Hospital de Jesus, D. F., D. F.
  - Hospital "Valentín Gómez Farías", Guadalajara, Jalisco
  - Instituto de Corazón de Querétaro, S.A. de C.V., Querétaro City, Querétaro
  - Cardioarritmias e Investigación, S.C., San Luis Potosí City, San Lusi Potosi
  - Hospital Cardiológica Aguascalientes, Aguascalientes
  - Cardioprevent, Durango
  - Hospital Angeles de Puebla, Puebla City
  - Hospital General de Puebla, Puebla City
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
- Poland (62):
  - Oddział Kardiologii z Zakładem Diagnostyki Kardiologicznej, Samodzielny Publiczny Zakład Opieki Zdrowotnej, Wojewódzki Szpital im. dr J. Biziela,, Bydgoszcz
  - NZOZ "Medicus" Jacek Kubica, Bydgoszcz
  - Wojewódzki Szpital Meijski im. Biziela, Oddział Kardiologii - SPZOZ, Bydgoszcz
  - Oddział Chorób Wewnętrzych i Kardiologii , ZOZ w Debicy, Dębica
  - Zakład Opieki Zdrowotnej Trójmiejskie Centrum Medyczne Sp. z o.o, Gdansk
  - Gabinet Kardiologiczny Medipuls, Gdynia
  - Gabinet Kardiologiczno-Internistyczny, Gdynia
  - Centrum Leczenia Chorób Cywilizacyjnych Oddz. Gdynia filla Fikakowo, Gdynia
  - NZOZ Medicus, Poradnia Kardiologiczna, Gliwice
  - Oddział Kardiologii i INK, SPZOZ nr 1, Gliwice
  - Mazowieckie Centrum Badań Klinicznych Iwona Czajkowska, Monika Śmietańska s.c., Grodzisk Mazowiecki
  - Publiczny Specjalistyczny Zaklad Opieki Zdrowotnej Oddzial Kardiologiczny, Inowrocław
  - Oddział Chorób Wewnętrznych i Farmakologii Klinicznej Samodzielny Publiczny Centralny Szpital Kliniczny im. Prof. Kornela Gibińskiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Szpital Specjalistyczny w Kościerzynie, Oddział Kardiologii, Kościerzyna
  - Oddział Kardiologii, Szpital Specjalistyczny im. J. Dietla, Krakow
  - "Klinika Choroby Wieńcowej Instytut Kardiologii, Collegium Medicum Uniwerytet Jagielloński, Krakow
  - Oddzial Chorób Wewnętrznych III Szpital Specjalistyczny im.Stefana Zeromskiego, SPZOZ w Krakowie, Krakow
  - Niepubliczny Zakład Opieki Zdrowotnej Specjalista Sp. z o.o., Kutno
  - Poradnia Kardiologiczna, Oddział Chorob Wewnetrznych Szpital Powiatowy w Limanowej, Limanowa
  - Niepubliczny Zakład Opieki Zdrowotnej POLIMEDICA, Lodz
  - All-Med Centrum Medyczne, Lodz
  - Oddział Internistyczno-Kardiologiczny Samodzielny Publiczny Zakład Opieki Zdrowotnej, Lubartów
  - "Oddzial Chorob Wewnetrznych i Kardiologii, Szpital Powiatowy im.Edmunda Biernackiego, Mielec
  - Oddział Kardiologii, Nowa Sól, Nowa Sól
  - "Oddział Kardiologiczno-Internistyczny, Olsztyn
  - "Oddział Kardiologiczny Publiczny Samodzielny ZOZ Wojewódzkie Centrum Medyczne, Opole
  - Specjalistyczny Zakład Opieki Zdrowotnej Poradnia lekarzy specjalistów "Jantar", Ostrów Wielkopolski
  - ZOZ w Oławie, Oddział Chorób Wewnętrznych, Oława
  - II Oddział Wewnętrzny Samodzielny Publiczny Zakład Opieki Zdrowotnej, Pabianice
  - "Samodzielny Szpital Wojewódzki im. Mikołaja Kopernika, Oddział Kardiologiczny, Piotrkow Trybunalski
  - Medyczne Centrum Hetmańska, Indywiualna Specjalistyczna Praktyka Lekarska, Dr n. med. Piotr Leszczyński, Poznan
  - Specjalistyczne Centrum Diagnostyczno-Lecznicze Bamberski Dwór, Poznan
  - Oddział Wewnetrzny I, Szpital Kolejowy im. dr med. Włodzimierza Roeslera, Pruszków
  - Samodzileny Publiczny Zakład Opieki Zdrowotnej w Puławach, Szpital Specjalistyczny, Puławy
  - Wojewódzki Szpital Zespolony, Oddział Kardiologiczny, Płock
  - Specjalistyczna Przychodnia Lekarska "Medikard", Płock
  - Zakład Hemodynamiki, Wojewódzki Szpital Specjalistyczny, Radom
  - "Oddział Kardiologii z Pododdziałem Ostrych Zespołów Wieńcowych i z Ośrodkiem Implantacji Rozruszników Serca,, Rzeszów
  - Oddział Kardiologii, SP ZZOZ Sandomierz, Sandomierz
  - Oddział Kardiologiczny Wojewódzki Szpital Specjalistyczy w Siedlcach, Siedlce
  - Oddział Kardiologii Samodzielny Publiczny Zakład Opieki Zdrowotnej w Sieradzu im. Kardynała Stefana Wyszyńskiego, Sieradz
  - "Oddział Kardiologii, Wojewódzki Szpital Zespolony w Skierniewicach, ", Skierniewice
  - NZOZ Przychodnia Zadebie, Przychodnia Kardiologiczna, Skierniewice
  - "Oddział Kardiologii Inwazyjnej i Angiologii z Pr. Hemodynamiki, Stalowa Wola
  - Szpital Specjalistyczny Św.Jana, Oddział Kardiologii,, Starogard Gdański
  - Indywidualna Specjalistyczna Praktyka Lekarska, Szczecin
  - Poradnia Kardiologiczna, Tarnów
  - Specjalistyczny Gabinet Lekarski Internistyczno-Kardiologiczny-Cardiology, Tarnów
  - Niepubliczny Zakład Opieki Zdrowotnej "Nasz Lekarz", Praktyka Grupowa Lekarzy Rodzinnych z Przychodnią Specjalistyczną, Torun
  - Oddział Kardiologii Wojewódzki Szpital Zespolony, Torun
  - Oddział Kardiologiczny Szpital Wolski im. dr Anny Gostyńskiej Samodzielny Publiczny Zakład Opieki Zdrowotnej, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny Akademii Medycznej w Warszawie, Warsaw
  - II Klinika Choroby Wieńcowej Instytutu Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala Wyszynskiego, Warsaw
  - Centrum Leczenia Chorób Cywilizacyjnych, Warsaw
  - Międzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - NZOZ Starówka, Warsaw
  - "Oddział Kardiologiczny Wałbrzyski Ośrodek Kardiologii Interwencyjnej Specjalityczny Szpital im. Dr Alfreda Sokołowskiego, Wałbrzych
  - Synexus SCM Sp.z o o., Wroclaw
  - Niepubliczny Zakład Opieki Zdrowotnej, Centrum Badań Klinicznych, Wroclaw
  - Osrodek Chorob Serca, Klinika Kardiologii 4 Wojskowy Szpital Kliniczny z Poliklinika - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Wroclaw
  - "Śląskie Centrum Chorób Serca, III Katedra i Oddział Kliniczny Kardiologii Śląskiego Uniwersytetu Medycznego, Zabrze
  - Oddział Kardiologiczny Szpital Wojewódzki im. Kardynała Stefana Wyszyńskiego, Łomża
- Research and Cardiovascular Corp., Ponce, Puerto Rico
- Romania (10):
  - Spitalul Clinic Judetean de Urgenta Bacau, Bacau
  - S.C. Duo Medical S.R.L., Bucharest
  - Centrul Medical SANA, Bucharest
  - Cardiomed SRL, Bucharest
  - Institutul Inimii "Niculae Stanicioiu", Cluj-Napoca
  - Cardiomed SRL, Craiova
  - Dr. C.I. Parhon Hospital, Iași
  - Clinical county Hospital, Sibiu
  - Institutul de Boli Cardiovasculare si Transplan Tg. Mures, Târgu Mureş
  - County Hospital, Timișoara
- Slovakia (11):
  - Novamed s.r.o., Banská Bystrica
  - Alian s.r.o., Bardejov
  - 5. Interna klinika LF UK, FNsP Bratislava, Nemocnica Ruzinov, Bratislava
  - Cardio D&R spol. s r.o., Košice
  - Kardiomed s.r.o., Lučenec
  - NZZ Kardiocentrum Nitra s.r.o., Nitra
  - MUDr. Tibor DURIS, CSc., s.r.o., Nové Zámky
  - Nemocnica s poliklinikou Považská Bystrica, Považská Bystrica
  - Fakultna Nemocnica Trencin, Trenčín
  - Žilpo s.r.o., Žilina
  - Medivasa s.r.o., Žilina
- Ukraine (7):
  - "Klinichne obyednannia shvydkoi medychnoi dopomogy, m. Dnipropetrovs'k,Dnipropetrovs'ka derzhavna medychna akademiya, kafedra gospital'noi terapii #2, Dnipropetrovsk
  - Oblasnyi klinichnyi kardiologichnyi dyspanser, m. Ivano-Frankivsk, Ivano-Frankivskyi derzhavnyi medychnyi universytet, kafedra terapii # 3, Ivano-Frankivsk
  - TOV "Kardiologichna klinika "Sertse i sudyny" m. Kyiv, Kyiv
  - Natsionalnyi naukovyi tsentr "Instytut kardiologii im. akad. M.D. Strazheska" AMN Ukrainy, m. Kyiv, viddilenia symptomatychnykh arterial'nykh gipertenziy, Kyiv
  - Natsionalnyi naukovyi tsentr "Instytut kardiologii im. akad. M.D. Strazheska", viddil reanimatsii ta intensyvnoi terapii, m. Kyiv, Kyiv
  - Komunal'na ustanova "Oblasnyi kardiologichnyi dyspanser", viddilenia intensyvnoi terapii, m. Zaporizhzhia, Zaporizhzhya
  - Kardioarytmologichnyi tsentr Zhytomyrs'koi oblasnoi klinichnoi likarni im. O.F. Gorbachevs'kogo, m. Zhytomyr, Zhytomyr

REFERENCES:
- [Derived] Vaduganathan M, Bhatt DL, Cryer BL, Liu Y, Hsieh WH, Doros G, Cohen M, Lanas A, Schnitzer TJ, Shook TL, Lapuerta P, Goldsmith MA, Laine L, Cannon CP; COGENT Investigators. Proton-Pump Inhibitors Reduce Gastrointestinal Events Regardless of Aspirin Dose in Patients Requiring Dual Antiplatelet Therapy. J Am Coll Cardiol. 2016 Apr 12;67(14):1661-71. doi: 10.1016/j.jacc.2015.12.068. Epub 2016 Mar 21. PMID 27012778
- [Derived] Bhatt DL, Cryer BL, Contant CF, Cohen M, Lanas A, Schnitzer TJ, Shook TL, Lapuerta P, Goldsmith MA, Laine L, Scirica BM, Murphy SA, Cannon CP; COGENT Investigators. Clopidogrel with or without omeprazole in coronary artery disease. N Engl J Med. 2010 Nov 11;363(20):1909-17. doi: 10.1056/NEJMoa1007964. Epub 2010 Oct 6. PMID 20925534